CLINICAL TRIAL: NCT04751851
Title: Determinants of Optimal Benzodiazepines Withdrawal in Adults With Hypnotic-dependent Insomnia: a Randomised Controlled Trial Evaluating Acceptance and Commitment Therapy in Telepsychology
Brief Title: Telepsychology for Benzodiazepines Withdrawal in Adults Suffering From Hypnotic-dependent Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale de Promotion des Connaissances sur le Sommeil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BENZOSTOP
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Chronic Insomnia; Hypnotic Dependence
Keywords: Benzodiazepines; Withdrawal; Acceptance and Commitment Therapy; Cognitive Behavioural Therapy; Telepsychology
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: The participants will be randomly divided into four arms :
  * Group A.1: Medium duration withdrawal programme with ACT
  * Group A.2: Long duration withdrawal programme with ACT
  * Group B.1: Medium duration withdrawal programme without ACT
  * Group B.2: Long duration withdrawal programme without ACT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- A.1: Medium duration withdrawal programme with ACT (Experimental): Medium duration withdrawal programme with Acceptance and Commitment Therapy
  Interventions: Behavioral: Medium duration withdrawal programme with ACT
- A.2: Long duration withdrawal programme with ACT (Experimental): Long duration withdrawal programme with Acceptance and Commitment Therapy
  Interventions: Behavioral: Long duration withdrawal programme with ACT
- B.1: Medium duration withdrawal programme without ACT (Active Comparator): Medium duration withdrawal programme without Acceptance and Commitment Therapy
  Interventions: Behavioral: Medium duration withdrawal programme without ACT
- B.2: Long duration withdrawal programme without ACT (Active Comparator): Long duration withdrawal programme without Acceptance and Commitment Therapy
  Interventions: Behavioral: Long duration withdrawal programme without ACT

INTERVENTIONS:
Behavioral: Medium duration withdrawal programme with ACT — * 10 interviews of withdrawal monitoring and psychological support during a taper programme of 6 weeks.
  * 8 individual weekly ACT sessions. The ACT programme includes mindfulness, acceptance and thoughts defusion exercises, identification of personal values and promotion of actions committed to these values. It also includes sleep restriction, a component of CBT for insomnia, used in this protocol to carry out committed-actions, according to the principles of ACT.
  Arms: A.1: Medium duration withdrawal programme with ACT
Behavioral: Long duration withdrawal programme with ACT — * 10 interviews of withdrawal monitoring and psychological support during a taper programme of 18 weeks.
  * 8 individual weekly ACT sessions. The ACT programme includes mindfulness, acceptance and thoughts defusion exercises, identification of personal values and promotion of actions committed to these values. It also includes sleep restriction, a component of CBT for insomnia, used in this protocol to carry out committed-actions, according to the principles of ACT.
  Arms: A.2: Long duration withdrawal programme with ACT
Behavioral: Medium duration withdrawal programme without ACT — 10 interviews of withdrawal monitoring and psychological support during a taper programme of 6 weeks.
  Arms: B.1: Medium duration withdrawal programme without ACT
Behavioral: Long duration withdrawal programme without ACT — 10 interviews of withdrawal monitoring and psychological support during a taper programme of 18 weeks.
  Arms: B.2: Long duration withdrawal programme without ACT

SUMMARY:
Long-term use of benzodiazepines is a long-standing problem, but the optimal withdrawal modalities are not known. The main objective of this study is to compare the effectiveness of a psychological support versus a psychotherapeutic intervention (Acceptance and Commitment Therapy, ACT) added to a withdrawal program on the reduction of benzodiazepines use in adults suffering from insomnia and hypnotic dependence.

DETAILED DESCRIPTION:
Benzodiazepines and related drugs (BZDs) are effective for insomnia and anxiety in the short term. After few months (four weeks regarding insomnia), the benefit/risk ratio is considerably reduced. Nevertheless, between 2 and 5% of the general population uses them for more than 6 months. Prescribing recommendations are unanimous concerning the short-term use of these substances, but do not specify the optimal ways of reducing doses in a withdrawal programme.

Many factors influence the success of withdrawal, including the duration of withdrawal (how quickly doses are reduced), the half-life of the substance, and number of psychological factors. Studies on BZD withdrawal show that, on average, spontaneous cessation of treatment is 5-10%, withdrawal success is 30-40% following brief intervention and 60-80% following Behavioral and Cognitive Therapy (CBT). These are few, and only one study has tested the efficacy of Acceptance and Commitment Therapy (ACT) for benzodiazepine withdrawal. ACT is a contextual behavioral therapy which aims to increase acceptance of the full range of inner experiences including negative thoughts, emotions and sensations, in order to promote values-driven behavior change, leading to an improved quality of life. ACT is notably effective for the treatment of anxiety disorders, depression, psychosis and chronic pain, and some studies have shown the effectiveness of ACT for insomnia.

This study is a four-arms randomized controlled intervention which aims to evaluate the addition to a taper program of an ACT intervention versus a psychological support on one hand, and the duration of withdrawal on the other hand, in patients suffering from hypnotic-dependent insomnia. The entire protocol will be remotely delivered, which no randomized controlled trial has so far evaluated for benzodiazepine withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* French speaker
* Had benzodiazepines and related drugs prescribed to improving sleep, for a minimum of 4 nights per week and for at least 6 months
* Pathological Benzodiazepine Dependence Questionnaire (BDEPQ) score (>34).
* Motivated to stop hypnotic treatment (score >5 on a 1 to 10 degrees VAS)
* Subjective complaints of difficulties initiating and/or maintaining sleep for a minimum of 3 nights per week and for at least 6 months, and 4) presence of marked distress or impaired daytime functioning (fatigue, impaired attention and/or concentration). Because hypnotic medications may mask an underlying insomnia problem, participants should meet these criteria either currently (while taking medication) or after previous attempts to discontinue the medication. These criteria are consistent with those for primary insomnia and hypnotic-dependent insomnia.
* Present the diagnoses of insomnia (307.42) and sedative, hypnotic and anxiolytic use disorder (304.10) from the DSM V.
* Having e-literacy (being familiar with emails, videoconferencing, online questionnaires and Internet use)

Exclusion Criteria:

* In acute treatment for psychological or psychiatric problems (e.g., current participation in psychotherapy)
* Be participating in a tapering BZD protocol, or similar
* Currently receiving an active prescription for any antipsychotic medication
* Using non-BZRA sedative-hypnotics for treating insomnia or related sleep problems (e.g., trazodone, quetiapine, tricyclic antidepressant, mirtazapine, diphenhydramine, dimenhydrinate)
* Met criteria for a substance use disorder in the last six months (other than nicotine and hypnotics)
* Use of alcohol or cannabis 3 or more nights a week for sleep problems
* Drinking more than 3 alcoholic beverages per day
* Presence of another untreated sleep disorder (e.g., obstructive sleep apnea or periodic limb movements during sleep)
* Presence of major depression or other severe unstabilized psychopathology (e.g., bipolar disorder, psychosis, panic disorder, generalized anxiety disorder, posttraumatic stress disorder, specific phobia, social phobia, or obsessive-compulsive disorder)
* Had a history of psychosis
* Currently suicidal
* Current crisis or with an illness for which the benzodiazepine were required at the time (e.g. acute pain)
* Presence of terminal illness (e.g. cancer, receiving palliative care)
* Unstable cardiovascular, respiratory or endocrinological diseases (clinical interview)
* Had a history of severe cognitive impairment, dementia, seizure disorder (epilepsy either in themselves or in their family), spinal injury
* Pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Proportion of participants having successfully stopped their benzodiazepine use | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Proportion of participants who successfully discontinue benzodiazepines (i.e., no benzodiazepine used for 2 weeks preceding assessment and negative on the urine test for BZD) at 4 weeks posttreatment, 6 months posttreatment, 12 months posttreatment and 24 months posttreatment. Successful discontinuation is defined as completion of the taper schedule without significant deviation and no use of benzodiazepine medications beyond "minimal Pro re nata. use" during the month following the zero-dose date. Minimal BZD use (not considered discontinuation failures): use of no more than 2 Pro Re Nata doses of medication (each not exceeding 0.5 mg diazepam) during the 2 weeks period starting at the zero-dose date. This criterion ensures that taking a minimal P.R.N. dose in extraordinary circumstances will not be considered discontinuation failures.

SECONDARY OUTCOMES:
Benzodiazepines use 1 | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Proportion of participants who were able to reduce the dose by 50% or more BZD (over the two weeks prior to the assessments)
Benzodiazepines use 2 | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Number of nights per week without BZD (over the two weeks preceding the assessments)
Benzodiazepines dependence | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Benzodiazepine Dependence Questionnaire (i.e. BDEPQ). This questionnaire evaluates the severity of BZD dependence via 30 items in 4 points, divided into 3 subscales: general dependence, pleasurable effect, perception of need.
Compliance | Change from 1 month post-treatment at 3 months, 12 months and 24 months post-treatment
  Significant deviation from the taper schedule (considered treatment failures) = failure to make a scheduled dose decrease for a 10 days period, or falling more than 14 days behind the allowed taper schedule dose for any consecutive three days period, or continued BZD use beyond 14 days from the scheduled zero-dose date.
Assessment of withdrawal symptoms | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Clinical Institute Withdrawal Assessment-B (CIWA-B) contains 20 5-point items designed to assess and monitor the type and severity of benzodiazepine-like withdrawal symptoms. The first three items (restlessness, tremor, and sweating) are rated by the treating physician, and the last 17 items are rated by the patient.
Sleep Improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  The severity of insomnia as measured by the Insomnia Severity Index (i.e., ISI). The ISI questionnaire assesses satisfaction, daily functioning and anxiety related to sleep problems with 7 5-point items.
Psychopathological symptoms improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Psychological distress as assessed by the Symptom Checklist 90, (i.e., SCL-90). The following 9 psychopathological dimensions are assessed by 90 5-point items: Somatization, Interpersonal sensitivity, Depression, Anxiety, Hostility and aggression, Obsessive-Compulsive, Phobic anxiety, Paranoid ideas, Psychoticism.
Quality of life improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Quality of life as measured by WHOQOL-26 (i.e., WHOQOL-BREF). This abbreviated form of the WHOQOL-100 assesses the following 4 dimensions: "physical health", "mental well-being", "social relationships" and "environment" by 26 5-point items.
Self-confidence in benzodiazepines reduction | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Self-confidence towards change in benzodiazepine use assessed by two questions: "How confident are you in stopping your benzodiazepines" (0% I can't stop my medication; 100% I feel able to stop my benzodiazepines) and "How confident are you in your ability to sleep without benzodiazepines" (0% I can't sleep without benzodiazepines; 100% I feel able to sleep without benzodiazepines).
Awareness improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Ability to be in contact with the present moment as measured by the Philadelphia Mindfulness Scale (i.e., MAAS) : 15 6-point items assess the capacity for mindfulness, i.e., the ability to pay attention without judgment to the present moment.
Psychological flexibility improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Psychological flexibility as measured by the Acceptance and Action Questionnaire (i.e., AAQ-II) : 10 7-point items assess the ability to not act solely to modify unpleasant psychological experiences.
Global ACT processes improvement | Change from baseline at 1 month, 3 months, 12 months and 24 months post-treatment
  Overall assessment of the 6 ACT processes as measured by the Comprehensive assessment of Acceptance and Commitment Therapy processes (i.e., CompACT). This 23-item questionnaire uses a 5-point scale to assess the following 6 dimensions, corresponding to the 6 ACT processes: Acceptance, Defusion, Contact with the present moment, Self as Context, Values, and Committed Actions.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Putois, MD, Ph.D, Principal Investigator — Lyon Neuroscience Research Centre, CNRS UMR 5292 - INSERM U1028 - Lyon 1 University, France; Laure Peter-Derex, MD, Ph.D, Principal Investigator — Lyon Neuroscience Research Centre, CNRS UMR 5292 - INSERM U1028 - Lyon 1 University, France
Locations (1):
- PROSOM, Lausanne, Switzerland